CLINICAL TRIAL: NCT06260696
Title: Assessing Health-Related Quality of Life and Willingness to Pay for Weight Management in Asia-Pacific by Gender
Acronym: ASPECT - APAC
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7626; U1111-1282-5512 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Normal weight: Adults with normal weight, recruited to complete self-administered online service
  Interventions: Other: No treatment is given
- Overweight: Adults with overweight, recruited to complete self-administered online service
  Interventions: Other: No treatment is given
- Obesity Class I: Adults with obesity class I, recruited to complete self-administered online service
  Interventions: Other: No treatment is given
- Obesity Class II: Adults with obesity class II, recruited to complete self-administered online service
  Interventions: Other: No treatment is given
- Obesity Class III: Adults with obesity class III, recruited to complete self-administered online service
  Interventions: Other: No treatment is given

INTERVENTIONS:
Other: No treatment is given — No treatment is given

SUMMARY:
The purpose of this survey is to collect information for scientific research and to identify the impact of overweight and obesity on health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Not currently pregnant
4. Does not participate in intense fitness or body building program
5. Weight loss not through illness or injury
6. Lives in South Korea, Australia, or India
7. BMI above or equal to 18 and associated weight class (Normal Weight or above) will be determined by a programmed calculation based on participant-reported height and weight.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Does not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults recruited to complete self-administered online service
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Score on IWQOL-Lite validated | At time of survey response (Day 1)
  Calculated score. Likert scale; 1=Never True, 5=Always True

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com